CLINICAL TRIAL: NCT07397312
Title: A Pilot Study to Test the Efficacy of a Commercial Toothpaste (Cosmetic Product)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Periotrap Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CosTP-001
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Periodontitis
Keywords: periodontitis; toothpaste
MeSH Terms: conditions — Periodontitis | interventions — Toothpastes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- toothpaste (Experimental)
  Interventions: Other: Toothpaste

INTERVENTIONS:
Other: Toothpaste — brushing teeth with toothpaste twice a day for and refrain from mouth rinsing after spitting out

SUMMARY:
This clinical multi-center, controlled, study will be carried out in volunteers with every 3- to 6-months professional tooth cleaning during their non-treatment period between 2 re-calls of a supportive periodontitis therapy regime. The efficacy of domestic oral hygiene by using a commercial dentifrice will be determined. Besides regularly used ingredients such as NaF and cleaning bodies the dentifrice contains a novel compound, which may be beneficial for the protection of an eubiotic oral microbiome. During the 3-month study period, participants will brush with their allocated study product twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Good general health with no clinically significant and relevant abnormalities of medical history.
* Absence of any condition that would impact on the subject's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.

At Screening (Visit 1):

* Participant with at least 16 natural, permanent teeth.
* A participant who gets regularly professional tooth cleaning in a frequence of once to twice yearly.
* Participant whose biofilm contains at least Porphyromonas gingivalis.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or a sponsor's employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who has any other clinical serious or unstable conditions (for example, cardiovascular diseases, diabetes, liver disorders, bleeding disorders, and kidney disorders) which could have affected study outcomes and/or participant safety.
* A participant who has a Plaque Control Record (PCR) > 35 %.
* A participant who plans to get pregnant during the study or is already pregnant (pregnancy testing) or breastfeeding.
* A participant who is known or suspected of intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who is unwilling or unable to comply with the lifestyle considerations.
* Participant who is a current smoker (more than 5 cigarettes per day).
* Participant who is using smokeless forms of tobacco (for example, chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).
* A participant who is diagnosed with xerostomia or is taking any medication that is causing xerostomia.
* A participant who has a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has a severe oral condition (for example, necrotizing gingivitis/periodontitis or oral or peri-oral ulceration) that could compromise study outcomes or the oral health of the participant/examiner if they participate in the study.
* A participant who has previously been enrolled in this study.

Medication exclusions at screening (Visit 1):

* A participant who is using any antibiotic medication within 3 months prior to inclusion or at any time during the study.
* A participant who is currently taking an anti-inflammatory or systemic medication (for example, immunosuppressants), which could affect plaque/gingival condition (for example, ibuprofen, aspirin, cyclosporin, phenytoin, calcium channel blockers) repeatedly for more than 3 consecutive days within study participation.

Periodontal and dental exclusions:

* A participant who has a formally untreated or not controlled periodontitis.
* A participant who has active caries that could compromise study outcomes or the oral health of the participant if they participate in the study.
* A participant who has an orthodontic appliance (bands, appliances, or fixed/ removable retainers except night guards).
* A participant who has any dental condition (for example, overcrowding) that could compromise study outcomes or the oral health of the participant if they participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy before and after 3 months of using newly developed microbiome-modulating toothpaste | From enrollment to the end of treatment at 12 weeks.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Dr. Hofmann, Bietigheim-Bissingen
  - Dr. T. Schütz, Borna
  - Dr. G. Jungbauer, Straubing